CLINICAL TRIAL: NCT01378754
Title: A DOSE RANGING STUDY TO EVALUATE THE EFFECTIVENESS OF FOSPROPOFOL (LUSEDRA®) FOR INDUCTION OF ANESTHESIA FOR OUTPATIENT UROLOGIC HYDRODILATION THERAPY
Brief Title: Evaluate The Effectiveness Of Fospropofol (Lusedra®) For Induction Of Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding before enrollment.
Sponsor: Grace Shih, MD (Other)
Responsible Party: Sponsor-Investigator, Grace Shih, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12588
Record Dates: First submitted 2011-06-08; First posted 2011-06-22 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Interstitial Cystitis
Keywords: hydrodilation; general anesthetic
MeSH Terms: conditions — Cystitis, Interstitial | interventions — fospropofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6.5 milligram per kilogram of Fospropofol (Lusedra®) (Experimental)
  Interventions: Drug: Fospropofol (Lusedra®) 6.5
- 10 milligram per kilogram of Fospropofol (Lusedra®) (Experimental)
  Interventions: Drug: Fospropofol (Lusedra®) 10
- 12 milligram per kilogram of Fospropofol (Lusedra®) (Experimental)
  Interventions: Drug: Fospropofol (Lusedra®) 12

INTERVENTIONS:
Drug: Fospropofol (Lusedra®) 6.5 — Group 1 will receive 6.5 milligram per kilogram of Fospropofol (Lusedra®) injection (IV).
  Arms: 6.5 milligram per kilogram of Fospropofol (Lusedra®)
Drug: Fospropofol (Lusedra®) 10 — Group 2 will receive 10 milligram per kilogram of Fospropofol (Lusedra®) injection (IV).
  Arms: 10 milligram per kilogram of Fospropofol (Lusedra®)
Drug: Fospropofol (Lusedra®) 12 — Group 3 will receive 12 milligram per kilogram of Fospropofol (Lusedra®) injection (IV).
  Arms: 12 milligram per kilogram of Fospropofol (Lusedra®)

SUMMARY:
Interstitial cystitis is a condition where a defect in the protective lining of the bladder causes the urinary symptoms such as urgency, frequency and pain/burning on urination. One way to help ease the symptoms of this disease is to fill the bladder full of water every 4 to 6 months.

Since this is a painful procedure an anesthesiologist will give you a drug that will make you unconscious for the procedure. General anesthesia can be given to you through an IV tube that is placed in a vein in your arm. There are only a few agents that induce sedation and these agents have certain disadvantages such as waking up slowly, low blood pressure, and pain at the injection site and a prolonged time to consciousness.

This study will be comparing doses of a new IV sedation induction agent drug to put you to sleep called fospropofol (Lusedra®).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients

  -> 18-65 years of age,
* weight 60-90 kg,
* with an American Society of Anesthesiologists (ASA) physical status of P1 to P3 are eligible for enrollment.
* Female patients of child bearing age will have a negative urine pregnancy test result and have used an acceptable method of birth control for >1 month prior to study enrollment.
* Patients will be NPO >6 hours and scheduled for outpatient urological hydrodilation under general anesthesia.
* Patients also will not be enrolled in another study or have received an experimental drug in the prior 30 days.

Exclusion criteria are:

* hypersensitivity or allergy to any anesthesia, opioids, benzodiazepines or any drugs used in the study, failure to meet NPO status or an abnormal, clinically significant ECG finding.
* Another exclusion is the presence of a difficult airway that would prevent use of the laryngeal mask airway (LMA) or successful LMA insertion.
* Women who are breast feeding would also be excluded from participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the differences in dose on the time to loss of consciousness and loss of reflex using the laryngeal mask airway (LMA). | 1 day
  To evaluate the use, dosing, efficacy and safety of fospropofol (Lusedra®) for the induction of general anesthesia using the laryngeal mask airway (LMA) in outpatient urology patients receiving hydrodilation therapy.

SECONDARY OUTCOMES:
To evaluate the difference in dose on blood pressure and heart rate using the laryngeal mask airway (LMA) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Grace Shih, MD, Principal Investigator — University of Kansas Medical Center